CLINICAL TRIAL: NCT02863198
Title: Endometrial Injury for Unexplained Infertility: Randomized Case-control Study
Brief Title: Endometrial Injury for Unexplained Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, khalid mohammed salama, director clinical research, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Khalid 3
Record Dates: First submitted 2016-08-04; First posted 2016-08-11 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-01

CONDITIONS: Infertility
Keywords: unexplained infertility; endometrial injury; pregnancy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- endometrial injury (Active Comparator): Endometrial injury was done only for patient of the study group. It was done on day 5, under complete aseptic conditions, no anesthesia, was given in most of cases. Endometrial local injury was performed on the posterior wall, midline, and 10-15 mm from the fundus using pipelle endometrial sampling (Pipelle).
  Interventions: Device: endometrial injury
- non endometrial injury (No Intervention): non endometrial injury was done only for patient of the control group

INTERVENTIONS:
Device: endometrial injury — Endometrial injury was done only for patient of the study group. It was done on day 5, under complete aseptic conditions, no anesthesia, was given in most of cases. Endometrial local injury was performed on the posterior wall, midline, and 10-15 mm from the fundus using pipelle endometrial sampling (Pipelle).
  Arms: endometrial injury

SUMMARY:
One hundred and twenty women with unexplained infertility were included in the study. Divided randomly into two groups:

Group I: (60 patients): (control group)

Group II (60 patients): (study group)

All the patients received (CC) and human menopausal gonadotropin. On day 5 of the cycle, Doppler examination was performed to all patients. Also on day 5, but only for group (II) patients, local endometrial injury was performed. Doppler studies was repeated, for all our patients, on the same day of prescribing human chorionic gonadotropin

DETAILED DESCRIPTION:
This randomized case-control study was performed at the Obstetrics and Gynecology Department of University Hospital, during the period between October 2013 till July 2015. One hundred and twenty women with unexplained infertility were included in the study.

Written, informed, consent, was taken from all women after explaining the nature and the aim of the study. The 120 patients were divided randomly into two groups (based on each alternate week referral to the clinic). All the patients received Clomiphene citrate (CC) and, Human menopausal gonadotrophin, according to the following protocol: Clomiphene Citrate (Clomiphene tablets, Clomiphene citrate 50 mg), 100 mg/day for 5 consecutive days, with therapy initiated on cycle day 3. Human menopausal gonadotrophin (Merional 75 international unit), was injected intra-muscularly, in a dose of 150 iu/day, on the days 3, 5, 7, 9 of the menstrual cycle. Serial transvaginal ultra sound was performed for all patients starting from day 10 and repeated every other day. Human menopausal gonadotrophin was continued daily, in the same dose, until follicles reached 18-22 mm. When the dominant follicles reached 18-22 mm, as measured by transvaginal ultrasound, human chorionic gonadotropin (5000 international unit) was injected intramuscularly, in a dose of 5,000 - 10,000 IU, and timed intercourse was advised, 36 h after human chorionic gonadotropin injection and the days after. Vaginal ultrasound was done about 60 h after human chorionic gonadotropin injection to confirm follicular rupture. On day 5 of the cycle, Doppler examination was performed to all patients. Also on day 5, but only for group II patients, local endometrial injury was performed. Doppler studies was repeated, for all our patients, on the same day of prescribing human chorionic gonadotropin.

Technique of trans vaginal ultrasound: Trans vaginal sonography examination was performed with patient in the lithotomy position using transvaginal transducer with color Doppler facility, a longitudinal view of the uterus was obtained then, the color Doppler mode was activated. The endometrial and subendometrial blood flow distribution pattern was determined by demonstrating pulsatile color signals in the sub endometrial and endometrial regions. Doppler sonography was performed on the vessels with the highest color intensity within the innermost endometrial and sub endometrial area. The insonation angle was kept at 0° to identify the course of the small spiral arteries. After confirming that waveforms were continuous, an average of three to five cardiac cycles were selected for calculation of resistance index (RI), pulsatility index (PI). The vessel with the lowest PI was considered for further statistical analysis. Uterine circulation was assessed simultaneously in each examination; bilateral uterine arteries were sampled lateral to the cervix near the internal os. Mean levels of both uterine RI and PI were used for analysis.on the day of human chorionic gonadotropin administration the endometrial thickness was measured, and reported. on the same day The endometrial pattern was evaluated and described as a multilayered or a non-multilayered endometrium. A trilaminar endometrium presented as a triple-line pattern in which hyperechogenic outer lines and a well-defined central echogenic line with hypoechogenic or black areas between these lines. A non trilaminar endometrium consisted of homogeneous endometrial patterns, characterized by either hyperechogenic or isoechoic endometrium.

Technique of endometrial injury: Endometrial injury was done only for patient of the study group. It was done on day 5, under complete aseptic conditions, no anesthesia, was given in most of cases. Endometrial local injury was performed on the posterior wall, midline, and 10-15 mm from the fundus using pipelle endometrial sampling (Pipelle).

ELIGIBILITY:
Inclusion Criteria:

* age Between 20 - 35 years
* Body mass index 18-29 kg/m2
* primary infertility for more than two years, and planning for IVF/intracytoplasmic sperm injection trial
* Normal ovulation confirmed by previous US
* Normal hormonal profile follicle stimulating hormone, luteinizing hormone, and prolactin, Antimullerian hormone (AMH) more than 1 ng/ml
* Normal hysterosalpingography
* Normal laparoscopic finding
* normal semen analysis, according to World Health Organization 2010

Exclusion Criteria:

* Absence of inclusion criteria
* History of previous laparotomy
* Patients with history which may suggest endometriosis
* Associated chronic medical conditions e.g. cardiac disease, diabetes, renal disease… etc.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: khalid M salama, Study Director — Benha University
Locations (1):
- Benha university hospitalا, Banhā, Alqalubia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maged AM, Al-Inany H, Salama KM, Souidan II, Abo Ragab HM, Elnassery N. Endometrial Scratch Injury Induces Higher Pregnancy Rate for Women With Unexplained Infertility Undergoing IUI With Ovarian Stimulation: A Randomized Controlled Trial. Reprod Sci. 2016 Feb;23(2):239-43. doi: 10.1177/1933719115602776. Epub 2015 Sep 3. PMID 26342054
- See also: infertility — http://bu.edu.eg

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endometrial Injury | Non Endometrial Injury
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endometrial Injury | Non Endometrial Injury | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 60 | 120
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 120
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Egypt | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Uterine Artery Pulsatility Index
Description: measurement of uterine artery pulsatility index at day of human chorionic gonadotropin administration.Pulsatility index is a measure of the variability of blood velocity in a vessel, and was calculated as the difference between the peak systolic and end diastolic velocities divided by the mean velocity during the cardiac cycle. Higher values are indicative of increased vascular resistance.
Time Frame: one week
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Endometrial Injury | Non Endometrial Injury
Number analyzed (Participants) | 60 | 60
index | 2.40 (0.23) | 2.35 (0.28)
Statistical Analysis 1: Comparison: Endometrial Injury vs Non Endometrial Injury; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — All included p-values are calculated from collected data and not threshold values for statical significance

2. Primary Outcome: Measurement of Uterine Artery Resistance Index
Description: measurement of uterine artery resistance index at day of human chorionic gonadotropin administration.it is an indicator of resistance of uterine artery to perfusion . In ultrasonography, it can be calculated from the peak systolic velocity and end diastolic velocity of blood flow and is calculated with the following formula: (peak systolic velocity - end diastolic velocity)/peak systolic velocity.lower values are better than higher values.
Time Frame: one week
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Endometrial Injury | Non Endometrial Injury
Number analyzed (Participants) | 60 | 60
index | 0.86 (0.04) | 0.85 (0.03)
Statistical Analysis 1: Comparison: Endometrial Injury vs Non Endometrial Injury; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — All included p-values are calculated from collected data and not threshold values for statical significance

3. Primary Outcome: Appearance of Sub Endometrial Blood Flow in All Patients
Description: Appearance of sub endometrial blood flow between patients of study and control groups on the day of human chorionic gonadotropin administration. subendometrial blood flow distribution pattern was determined by demonstrating pulsatile color signals in the sub endometrial area.The number of patients demonstrating subendometrial blood flow distribution pattern are collected .
Time Frame: one week
Measure: Number; unit: participants
Arm/Group | Endometrial Injury | Non Endometrial Injury
Number analyzed (Participants) | 60 | 60
participants | 33 | 12
Statistical Analysis 1: Comparison: Endometrial Injury vs Non Endometrial Injury; Test type: Superiority or Other; p < 0.05, Chi-squared — All included p-values are calculated from collected data and not threshold values for statical significance

4. Primary Outcome: Spiral Artery Pulsatility Indices in All Patients
Description: Spiral artery Doppler pulsatility indices between study and control groups on the day of human chorionic gonadotropin administration.Pulsatility index is a measure of the variability of blood velocity in a vessel, and was calculated as the difference between the peak systolic and end diastolic velocities divided by the mean velocity during the cardiac cycle. Higher values are indicative of increased vascular resistance
Time Frame: one week
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Endometrial Injury | Non Endometrial Injury
Number analyzed (Participants) | 60 | 60
index | 1.19 (0.246) | 1.01 (0.25)
Statistical Analysis 1: Comparison: Endometrial Injury vs Non Endometrial Injury; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — All included p-values are calculated from collected data and not threshold values for statical significance

5. Primary Outcome: Spiral Artery Doppler Resistance Indices in All Patients
Description: Spiral artery Doppler resistance indices between study and control groups on the day of human chorionic gonadotropin administration.it is an indicator of resistance of Spiral artery to perfusion . In ultrasonography,it can be calculated from the peak systolic velocity and end diastolic velocity of blood flow and is calculated with the following formula: (peak systolic velocity - end diastolic velocity)/peak systolic velocity.lower values are better than higher values.
Time Frame: one week
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Endometrial Injury | Non Endometrial Injury
Number analyzed (Participants) | 60 | 60
index | 0.62 (0.06) | 0.66 (0.04)
Statistical Analysis 1: Comparison: Endometrial Injury vs Non Endometrial Injury; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — All included p-values are calculated from collected data and not threshold values for statical significance

6. Secondary Outcome: Pregnancy Rate Between the Study and the Control Group
Description: detection of serum pregnancy tests for both groups( study and the control group)
Time Frame: 3 weeks
Measure: Number; unit: participants
Arm/Group | Endometrial Injury | Non Endometrial Injury
Number analyzed (Participants) | 60 | 60
participants | 11 | 4
Statistical Analysis 1: Comparison: Endometrial Injury vs Non Endometrial Injury; Test type: Superiority or Other; p < 0.05, Chi-squared — All included p-values are calculated from collected data and not threshold values for statical significance

ADVERSE EVENTS:
Arm/Group | Endometrial Injury | Non Endometrial Injury
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

LIMITATIONS AND CAVEATS:
No limitation or caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes